CLINICAL TRIAL: NCT00912561
Title: Effects of Intense Aerobic Exercise on the Cerebrovascular Reserve Capacity in Patients With Hemodynamically Relevant Intra- and Extracranial Stenoses
Acronym: Exercise
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruiting
Sponsor: Gerhard Jan Jungehuelsing (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Gerhard Jan Jungehuelsing, MD, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCBF-Exercise; EA4/106/08
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Stenosis
Keywords: chronic brain ischaemia; stroke prevention; exercise; physical training; Chronic, extra- or intracranial stenoses of brain supplying arteries
MeSH Terms: conditions — Constriction, Pathologic; Motor Activity; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sedentary (No Intervention): patients who train after an 8 week observational period
- patients who train immediately after enrollment (Active Comparator): patients who train immediately after enrollment
  Interventions: Behavioral: Intense aerobic exercise

INTERVENTIONS:
Behavioral: Intense aerobic exercise — 3 Units (of at least 30 minutes) of intense aerobic exercise per week for 8 weeks
  Arms: patients who train immediately after enrollment

SUMMARY:
The purpose of this trial is to study the improvement of cerebral hemodynamics in high risk stroke patients with impaired Cerebrovascular Reserve (CVR) due to high grade stenosis of the internal carotid (ICA) or middle cerebral artery (MCA) by Intense Aerobic Exercise (IAEx).

DETAILED DESCRIPTION:
The primary objective: Intense aerobic exercise (24/8 weeks) improves CVR > 20% measured by Transcranial Doppler (TCD) in patients with hemodynamic relevant intra- or extracranial stenoses by enhanced cerebral arterio- and angiogenesis.

Secondary objectives:

Intense aerobic exercise (24/8 weeks) leads to:

* an increase of Endothelial progenitor cell counts (EPCs)
* qualitative and quantitative changes of endothelial markers and cytokines representing the inflammatory activity of atherosclerosis and neovascularisation
* an improvement in cognitive performance and quality of life (QoL)
* changes of the mean vessel size and of cerebral perfusion

ELIGIBILITY:
Inclusion Criteria:

* high-grade stenosis of the intra- or extracranial ICA or the MCA with ipsilateral impairment of the CVR capacity measured by TCD

Exclusion Criteria:

* continuous physical activity ≥ 60 min/week within the last 3 months
* cerebral bleeding or ischaemic stroke < 3 months
* contraindications for spiro-ergometry, IAEx, or MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
change of cerebrovascular reserve capacity | immediately after intervention of 8 weeks, 3 months, 6 months, 12 months Follow up

SECONDARY OUTCOMES:
Endothelial Progenitor Cells, cyto- and chemokines | after intervention of 8 weeks, 3 months, 6 months, 12 months Follow up
Neuropsychological Testing/ Quality of life | immediately after intervention of 8 weeks, 3 months, 6 months, 12 months Follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Stroke Research Berlin, Neurology, Charité Campus Benjamin Franklin, Berlin, Germany